CLINICAL TRIAL: NCT01579565
Title: A Phase 3 Randomized, Double-Masked, Placebo-Controlled Study of the Pharmacokinetics of OMS302 and the Effect of OMS302 on Intraoperative Pupil Diameter and Early Postoperative Pain in Subjects Undergoing Intraocular Lens Replacement With Phacoemulsification
Brief Title: Safety, Efficacy and Pharmacokinetics of OMS302 in Subjects Undergoing Intraocular Lens Replacement With Phacoemulsification
Acronym: OMS302-ILR-004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS302-ILR-004
Record Dates: First submitted 2012-04-13; First posted 2012-04-18 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2014-08

CONDITIONS: Intraocular Lens Replacement
Keywords: cataract; lens replacement
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMS302 (Experimental): OMS302 diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Interventions: Drug: OMS302
- Placebo (Placebo Comparator): Placebo diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMS302 — OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL solution containing 60.75 millimolar (mM) phenylephrine hydrochloride (HCl) and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product is added to a 500 mL bottle of commercially available balanced saline salt (BSS) through a syringe filter. This will achieve 4.0 mL of the drug product in a 500 mL bottle of BSS.
  Arms: OMS302
Drug: Placebo — Placebo drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL solution containing 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product is added to a 500 mL bottle of commercially available BSS through a syringe filter. This will achieve 4.0 mL of the drug product in a 500 mL bottle of BSS.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, efficacy and pharmacokinetics of OMS302 (the study drug) for maintaining intraoperative mydriasis and preventing post operative pain in individuals undergoing Intraocular Lens Replacement (ILR) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Competent and willing to voluntarily provide informed consent
* 18 years of age or older
* In good general health needing to undergo cataract extraction or lens extraction with lens replacement surgery in one eye, under topical anesthesia

Exclusion Criteria:

* No allergies to the medications and/or the active ingredients of any of the study medications
* No medications with the same activities of the active ingredients in OMS302 for defined time intervals prior to and after surgery
* No other significant eye injuries, eye conditions or general medical conditions likely to interfere with the evaluation of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (14):
- United States (13):
  - Chandler, Arizona
  - Los Angeles, California
  - Fort Myers, Florida
  - Boston, Massachusetts
  - St Louis, Missouri
  - Washington, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Goodlettsville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
- Zwolle, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- OMS302: OMS302 diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  OMS302: OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 60.75 millimolar (mM) phenylephrine hydrochloride (HCl) and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available balanced saline solution (BSS) through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
- Placebo: Placebo diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Placebo: Placebo drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
Period: Randomized
Arm/Group | OMS302 | Placebo
Started | 207 | 209
Completed | 202 | 204
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — inadequate preoperative pupil dilation | 0 | 1
Not completed — prohibited preoperative eating | 1 | 0
Not completed — prohibited preoperative medication | 0 | 1
Period: Treated
Arm/Group | OMS302 | Placebo
Started | 202 | 204
Completed | 200 | 201
Not Completed | 2 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — declined to return for final visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- OMS302: OMS302 diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  OMS302: OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 60.75 mM phenylephrine HCl and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS solution through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
- Placebo: Placebo diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Placebo: Placebo drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS solution through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
- Total: Total of all reporting groups
Arm/Group | OMS302 | Placebo | Total
Number analyzed (Participants) | 202 | 204 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.2) | 67.5 (10.6) | 68.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 126 | 243
  Male | 85 | 78 | 163

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve Analysis of Change-from-Baseline in Pupil Diameter (mm) During Surgery
Description: The co-primary analysis of the change in pupil diameter based on the mean area under the curve (AUC) pupil diameter change from baseline. First, the AUC of the pupil diameter from surgical baseline to wound closure was calculated using the trapezoidal rule. Second, the mean AUC was obtained by dividing the AUC by the total time of surgery. Third, the mean AUC of change from baseline was calculated by subtracting the baseline pupil diameter from the mean AUC.
Time Frame: From surgery baseline (pre-incision) through surgery end (time of cortical clean-up/wound closure)
Population: Subjects with interpretable video images obtained during intraocular lens replacement (ILR) procedure.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- OMS302: OMS302 diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  OMS302: OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 60.75 mM phenylephrine HCl and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 195 | 200
mm | 0.1 (0.43) | -0.5 (0.57)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — p-value based on the generalized Cochran-Mantel-Haenszel (CMH) test stratified by the randomization strata; CMH-weighted mean difference (OMS302 - Placebo) is adjusted for the randomization strata; Mean Difference (Final Values) = 0.590, 95% CI [0.494 to 0.686], Standard Error of Mean 0.049

2. Primary Outcome: Mean Area Under the Curve Analysis of Ocular Pain VAS Score Within 12 Hours Postoperatively
Description: The co-primary analysis of the ocular pain VAS (where 0 = no pain and 100 = worst possible pain) based on the mean area under the curve (AUC). The AUC of the ocular pain VAS during 12 hours postoperatively was calculated by the trapezoidal rule in which the hour 11 was used to represent the time-point 10-12 hour. The mean AUC was defined as the AUC divided by the number of hours with ocular pain VAS results during the first 12 hours postoperatively.
Time Frame: 12 hours postoperatively
Population: Subjects with scores at time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 202 | 202
units on a scale | 4.3 (8.75) | 8.9 (15.19)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — p-value is based on the generalized CMH test stratified by the randomization strata; CMH-weighted mean difference (OMS302 - Placebo) is adjusted for the randomization strata; Mean Difference (Final Values) = -4.580, 95% CI [-6.917 to -2.244], Standard Error of Mean 1.192

3. Secondary Outcome: Pupil Diameter Greater Than or Equal to 6 mm at Completion of Cortical Clean up
Description: The number of subjects with pupil diameter of at least 6 mm at the completion of cortical clean up summarized by treatment arm. The last pupil diameter was used if not available at completion of cortical clean up.
Time Frame: at time of cortical clean-up (i.e., end of surgical procedure)
Population: Subjects with interpretable video images obtained during ILR procedure.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 195 | 200
participants | 187 | 154
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0001, Chi-squared — Chi-square test

4. Secondary Outcome: Pupil Diameter Less Than 6 mm Anytime During Surgery
Description: The number of subjects with pupil diameter less than 6 mm at any time during surgery summarized by treatment arm.
Time Frame: Intraoperative
Population: Subjects with interpretable video images obtained during ILR procedure.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 195 | 200
participants | 18 | 76
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0001, Chi-squared — Chi-square test

5. Secondary Outcome: Moderate-to-Severe Pain (VAS Greater Than or Equal to 40) at Any Time Point During 12 Hours Postoperatively
Description: The number of subjects with moderate -to-severe pain (VAS greater than or equal to 40) at any time point during 12 hours postoperatively summarized by treatment arm.
Time Frame: 12 hours postoperatively
Population: Subjects with VAS scores at time points.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 202 | 202
participants | 16 | 27
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0760, Chi-squared — Chi-square test

6. Secondary Outcome: Ocular Pain-Free (VAS Equal to 0) at All Time Points During 12 Hours Postoperatively
Description: The number of subjects who report ocular pain-free status (VAS equal to 0) at all time points during 12 hours postoperatively summarized by treatment arm. Subjects with missing VAS scores during the 12 hours postoperatively were considered as not being pain-free.
Time Frame: 12 hours postoperatively
Population: Subjects with scores at time points.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 202 | 202
participants | 56 | 41
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0806, Chi-squared — Chi-square test

7. Secondary Outcome: Ocular Pain VAS Score on Day 1
Description: VAS pain scores (where 0 = no pain and 100 = worst possible pain) after the day of surgery summarized by treatment arm and time point.
Time Frame: One day postoperatively
Population: Subjects with score at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 202 | 204
units on a scale | 5.8 (13.1) | 12.2 (20.1)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — Generalized CMH test stratified by randomization strata

8. Secondary Outcome: Ocular Symptoms Using Numerical Rating System (NRS) - Photophobia 6 Hours Post-Surgery
Description: Photophobia outcomes based on Ocular Pain and Symptoms Numerical Ordinal Scale (Numerical Rating System - NRS) at each time point.
Time Frame: Six hours postoperatively
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 200 | 202
participants
  None | 140 | 128
  Mild | 51 | 58
  Moderate | 8 | 13
  Severe | 1 | 3
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.3923, Cochran-Mantel-Haenszel — Treatment comparisons are based on Cochran-Mantel-Haenszel test adjusting for the randomization strata

9. Secondary Outcome: Ocular Symptoms Using Numerical Rating System (NRS) - Photophobia 1 Day Post-Surgery
Description: as for outcome 8
Time Frame: One day postoperatively
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 202 | 204
participants
  None | 119 | 95
  Mild | 63 | 63
  Moderate | 16 | 37
  Severe | 4 | 9
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0060, Cochran-Mantel-Haenszel — Treatment comparisons are based on Cochran-Mantel-Haenszel test adjusting for the randomization strata

10. Secondary Outcome: Postoperative Ocular Inflammation - Mean Summed Ocular Inflammation Score (SOIS) on Day 1
Description: Postoperative inflammation as measured using the Summed Ocular Inflammation Score (SOIS), summarized by treatment arm and time point. Ocular inflammation was evaluated by measuring the anterior chamber cell count and flare using a slit lamp biomicroscope. SOIS was calculated by adding the average of subject's anterior chamber cells and flare grades. The minimum SOIS was 0 (indicating absence of inflammation), whereas the maximum SOIS was 8.
  Grading was as follows:
  Anterior Chamber Cells: Grade None = 0/no cells; Grade Mild = +1/1-5 cells; Grade Moderate = +2/6-15 cells; Grade Severe = +3/16-30 cells; Grade Very Severe = +4/>30 cells.
  Anterior Chamber Flare: Grade None = 0/no Tyndall effect; Grade Mild = +1/barely discernable Tyndall effect; Grade Moderate = +2/moderately intense Tyndall beam in anterior chamber; Grade Severe = +3/severely intense Tyndall beam; Grade Very Severe = +4/very severely intense Tyndall beam with a white and milky appearance to the aqueous
Time Frame: One day postoperatively
Population: Subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 202 | 204
units on a scale | 2.8 (1.0) | 2.9 (1.3)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.3286, Cochran-Mantel-Haenszel — Treatment comparisons are based on generalized CMH test stratified by randomization strata

11. Secondary Outcome: Postoperative Best Corrected Visual Acuity (BVCA) on Day 1
Description: Best Corrected Visual Acuity (BCVA) summarized by the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity log score. The reason for missing scores (e.g., subject could not read enough letters to obtain a score or refraction was not completed) was also summarized. For subjects without a score due to inability to read the ETDRS chart, the log score was imputed as 1.6 for the purpose of treatment comparisons. Subjects without a score because the manifest refraction was not completed were excluded from the analysis.
Time Frame: One day postoperatively
Population: Subjects with score at time point.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 201 | 203
Log score | 0.1 (0.20) | 0.1 (0.18)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.2361, Wilcoxon rank-sum test — Treatment comparisons based on Wilcoxon rank-sum test stratified by randomization strata

12. Secondary Outcome: Systemic Pharmacokinetics (PK) of OMS302
Description: Systemic pharmacokinetics (PK) of phenylephrine (PE) and ketorolac (KE) were performed in a subset of subjects. Descriptive summary statistics for area-under-the-serum-concentration-time curve (AUC), maximum concentration (Cmax), time to Cmax (Tmax), and terminal phase half-life (t1/2) were to be generated if measured plasma concentrations were adequate for analysis. Descriptive statistics for pharmacokinetics were not performed as detected concentrations were low and insufficient for analysis.
Time Frame: 24 hours
Population: Subset of subjects randomized to OMS302 treatment.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 14 | 12
participants
  Subjects with detectable PE | 1 | 0
  Subjects with detectable KE | 10 | 1

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Placebo: Placebo diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Placebo: Placebo drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL solution containing 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product is added to a 500 mL bottle of commercially available BSS through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
Arm/Group | OMS302 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/202 | 2/204
Other Adverse Events (participants affected / at risk) | 118/202 | 143/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMS302 (N=202) | Placebo (N=204)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OMS302 (N=202) | Placebo (N=204)
Eye pain (Eye disorders) | 34 | 76
Headache (Nervous system disorders) | 21 | 24
Posterior capsule opafication (Eye disorders) | 17 | 14
Anterior chamber inflammation (Eye disorders) | 17 | 13
Ocular discomfort (Eye disorders) | 10 | 15
Vision blurred (Eye disorders) | 5 | 16
Conjunctival hyperaemia (Eye disorders) | 10 | 10
Photophobia (Eye disorders) | 4 | 13
Intraocular pressure increased (Investigations) | 12 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agreed not to publish or otherwise to disclose Study data without prior written consent from the sponsor for a period of 24 months following Study completion or until data are published in a combined publication (whichever occurs first). The sponsor can review communications containing results prior to public release and embargo those communications for a period that is no longer than 60 days from the date of receipt of the non-public communication. The sponsor cannot extend the embargo.